CLINICAL TRIAL: NCT00417612
Title: The Role of Parathyroid Hormone in the Pathogenesis of Skeletal Disease in X-linked Hypophosphatemic Rickets (XLH)
Brief Title: Effectiveness of Paricalcitol in Reducing Parathyroid Hormone (PTH) Levels in X-linked Hypophosphatemic Rickets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Thomas Carpenter, Professor of Pediatrics, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0607001636; P50AR054086 (NIH); 1P50AR054086-01 (NIH)
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Hypophosphatemia, Familial; Hyperparathyroidism
Keywords: Rickets, Hypophosphatemia; Rickets, Vitamin D-Resistant; Rickets, X-linked hypophosphatemic
MeSH Terms: conditions — Hypophosphatemia, Familial; Hyperparathyroidism; Rickets; Hypophosphatemia; Rickets, Hypophosphatemic; Familial Hypophosphatemic Rickets | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants given active drug, paricalcitol (Zemplar), in effort to reduce PTH level
  Interventions: Drug: Paricalcitol
- 2 (Placebo Comparator): Participants given placebo capsule to match for comparison
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol given first as a dose of 2 capsules once per day. Dose titration as needed per biochemical results at outpatient visits.
  Other Names: Zemplar
  Arms: 1
Other: Placebo — Placebo sugar pill
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness of paricalcitol, a form of synthetic vitamin D, in lowering parathyroid hormone (PTH) levels and reducing disease symptoms in children and adults with X-linked hypophosphatemic (XLH) rickets.

DETAILED DESCRIPTION:
XLH rickets is a rare inherited disorder in which the bones become painfully soft and bend easily because of a phosphate deficiency. This genetic defect causes the kidneys to allow excretion of an inappropriately high amount of phosphate into the urine. The kidneys are also unable to convert vitamin D into a form usable by the body, resulting in inadequate amounts of active vitamin D. Because vitamin D is needed to absorb calcium and phosphate from the intestine, this deficiency further reduces phosphate levels. Without the sufficient phosphate needed for normal bone growth, individuals with XLH rickets typically develop skeletal malformations, bone pain, and abnormally bowed legs. Hyperparathyroidism, a condition in which the parathyroid glands excrete excess amounts of PTH, also occurs frequently in individuals with XLH rickets, and may play a significant role in the skeletal complications associated with XLH rickets. The purpose of this study is to determine the effectiveness of paricalcitol in lowering PTH levels and reducing disease symptoms in individuals with XLH rickets.

This study will last 12 months. Participants will be randomly assigned to receive either paricalcitol or placebo, taken in the form of two pills daily for the duration of the study. During a baseline 3-day inpatient hospital stay, participants will undergo a physical exam, a cardiac ultrasound, a bone scan, blood collection, and a radiographic skeletal survey. The skeletal survey will include x-rays of various body parts. Participants who are 18 years or younger will not undergo the radiographic skeletal survey. Study visits for all participants will occur every 2 months until the end of the study. These visits will include a physical exam, review of disease symptoms, blood and urine collection, and a check of medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of XLH rickets
* Fasting serum calcium of 10.7 mg/dl or less
* Fasting PTH greater than 40 nleq/ml and less than 120 nleq/ml in the mid-molecule PTH assay at screening (upper limit of normal is 25 nleq/ml)
* Willing and able to participate in the trial
* Taking stable dose of standard therapy for XLH rickets for at least 2 months prior to study entry
* Concomitant therapy for XLH rickets will not be an exclusion criteria
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Concomitant kidney failure (estimated creatinine clearance less than 60 cc/min or serum creatinine greater than 1.5 mg/dl)
* Serum 25-hydroxy vitamin D less than 20 ng/ml. Participants meeting this criterion will receive vitamin D3 supplementation for 3 months and then be rescreened.
* Unable to comply with protocol and appropriate follow-up visits
* Treatment with agents that may affect skeletal metabolism, such as glucocorticoids and anticonvulsants

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O. Carpenter, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Brown AJ, Dusso AS, Slatopolsky E. Vitamin D analogues for secondary hyperparathyroidism. Nephrol Dial Transplant. 2002;17 Suppl 10:10-9. doi: 10.1093/ndt/17.suppl_10.10. PMID 12386264
- [Background] McElduff A, Posen S. Parathyroid hormone sensitivity in familial X-linked hypophosphatemic rickets. J Clin Endocrinol Metab. 1989 Aug;69(2):386-9. doi: 10.1210/jcem-69-2-386. PMID 2753981
- [Derived] Carpenter TO, Olear EA, Zhang JH, Ellis BK, Simpson CA, Cheng D, Gundberg CM, Insogna KL. Effect of paricalcitol on circulating parathyroid hormone in X-linked hypophosphatemia: a randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2014 Sep;99(9):3103-11. doi: 10.1210/jc.2014-2017. Epub 2014 Jul 16. PMID 25029424

RESULTS

PARTICIPANT FLOW:
Groups:
- Paricalcitol (Active Drug): Participants given active drug, paricalcitol (Zemplar), in effort to reduce Parathyroid Hormone (PTH) level
  Paricalcitol: Paricalcitol given first as a dose of 2 capsules once per day. Dose titration as needed per biochemical results at outpatient visits.
- Placebo: Participants given placebo capsule to match for comparison
  Placebo: Placebo sugar pill
Period: Overall Study
Arm/Group | Paricalcitol (Active Drug) | Placebo
Started | 22 | 11
Completed | 19 | 8
Not Completed | 3 | 3
Not completed — Errant diagnosis | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paricalcitol (Active Drug): Participants given active drug, paricalcitol (Zemplar), in effort to reduce PTH level
  Paricalcitol: Paricalcitol given first as a dose of 2 capsules once per day. Dose titration as needed per biochemical results at outpatient visits.
- Total: Total of all reporting groups
Arm/Group | Paricalcitol (Active Drug) | Placebo | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Parathyroid Hormone (PTHauc) Measurement
Description: Mean area under the curve for parathyroid hormone levels (PTHauc) sampled during a 26 hour study period, for Paricalcitol (Active Drug) and Placebo groups at Baseline and Month 12 .
Time Frame: Measured at baseline and Month 12
Measure: Mean (Standard Deviation); unit: nlEq*26hr/ml
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
nlEq*26hr/ml
  Baseline | 1223 (426) | 1449 (865)
  Month 12 | 987 (372) | 1616 (945)
Statistical Analysis 1: Comparison: Paricalcitol (Active Drug) vs Placebo; Test type: Superiority or Other; p = 0.007, ANOVA

2. Secondary Outcome: Static Parameters of Serum Alkaline Phosphatase at Baseline and 1 Year for Paricalcitol and Placebo Arms.
Time Frame: Measured at baseline and Month 12
Population: Alkaline phosphatase activity was analyzed separately for children (less than 18 years of age) and adults as values varied considerably between these two groups. In other outcome measure modules the paricalcitol group is comprised of 19 participants analyzed which includes adults and children. In this module, the children (2) are their own arm.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Paricalcitol (Children Ages 9-17): Pediatric patients ages 9-17 given paricalcitol
Arm/Group | Paricalcitol (Active Drug) | Placebo | Paricalcitol (Children Ages 9-17)
Number analyzed (Participants) | 17 | 8 | 2
mg/dl
  Serum Alkaline Phosphatase (Baseline) | 141 (96) | 96 (28) | 354 (2)
  Serum Alkaline Phosphatase (1 Year) | 112 (70) | 98 (34) | 402 (211)

3. Secondary Outcome: Serum Calcium
Time Frame: Measured at baseline and Month 12
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
mg/dl
  Serum Calcium (Baseline) | 9.2 (0.5) | 9.3 (0.5)
  Serum Calcium (1 Year) | 9.4 (0.5) | 9.3 (0.5)

4. Secondary Outcome: Bone Scan Severity Score
Description: 99-Tc-methylenediphosphonate bone scans were completed and analyzed using the following scale*: Bone scan severity scale with minimum score of 0 and maximum score of 4 (0 is no disease and 4 is greatest severity of disease).
  Appearance of lumbar spine and the sacroiliac region were used as internal references to which all suspected lesions were compared, and scored as follows:
  grade 0, normal scan without suspicious lesions grade 1, lesion(s) less intense than normal lumbar spine grade 2, lesion(s) similar in intensity to normal lumbar spine grade 3, lesions more intense than normal lumbar spine but similar to the normal sacroiliac region grade 4, lesions more intense than the normal sacroiliac region.
  *devised by nuclear medicine radiologist at Yale New Haven Hospital
Time Frame: Measured at baseline and Month 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
units on a scale
  Baseline Scan Score | 2.18 (1.19) | 2.00 (1.51)
  12 Month Scan Score | 1.76 (1.25) | 2.12 (1.55)

5. Secondary Outcome: Percent Change in Urinary Calcium Excretion From Baseline to 1 Year
Description: Percent change in daily urinary calcium excretion, which is calculated the measurements of the calcium in the subject's 24-hr urine collections done at baseline and at the 1 year timepoints
Time Frame: Measured at baseline and Month 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
percent change | 253 (388) | 9 (36)

6. Secondary Outcome: Serum Intact Fibroblast Growth Factor 23 (FGF23)
Time Frame: Measured at baseline and Month 12
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
pg/ml
  Serum Intact FGF23 (Baseline) | 120 [72 to 203] | 93 [46 to 188]
  Serum Intact FGF23 (1 Year) | 244 [145 to 411] | 104 [47 to 227]

7. Secondary Outcome: Serum 1,25 (OH)2D
Time Frame: Measured at baseline and Month 12
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
pg/ml
  Serum 1,25(OH)2D (Baseline) | 51 (18) | 47 (9)
  Serum 1,25 (OH)2D (1 Year) | 52 (17) | 46 (14)

8. Primary Outcome: Area Under the Curve for Parathyroid Hormone (PTH; Percentage Decrease)
Description: Mean PTHauc (% decrease) for Paricalcitol (Active Drug) and Placebo from Baseline to Month 12.
Time Frame: Measured at baseline and Month 12
Measure: Number; unit: participants
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
participants
  20-29% | 5 | 1
  30-39% | 1 | 1
  >/= 40% | 3 | 0

9. Primary Outcome: Reduction of Parathyroid Hormone Area Under the Curve (PTHauc) of 20% or Greater
Description: Clinically significant reduction of Mean PTHauc (% decrease >/= 20) for Paricalcitol (Active Drug) and Placebo from Baseline to Month 12.
Time Frame: Measured at baseline and Month 12
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol (Active Drug) | Placebo
Number analyzed (Participants) | 19 | 8
percentage of participants | 53 | 25

ADVERSE EVENTS:
Arm/Group | Paricalcitol (Active Drug) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/11
Other Adverse Events (participants affected / at risk) | 2/22 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (Active Drug) (N=22) | Placebo (N=11)
Elevated Serum Creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No